CLINICAL TRIAL: NCT06980662
Title: The Effect of Laughter Yoga in Beta Thalassaemia Major Patients: a Randomised Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Zeynep Bozan, STUDENT, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-SBE-ZB-01
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Beta Thalassemia Major; Thalassemia Majors (Beta-Thalassemia Major)
Keywords: Nursing, Fatigue, Depression-Anxiety-Stress and Sleep quality; fatigue
MeSH Terms: conditions — beta-Thalassemia; Fatigue; Sleep Initiation and Maintenance Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Two groups with a laughter yoga therapy control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group of patients will receive laughter yoga. Laughter yoga is a type of complementary therapy that also includes some other components, including light physical exercises. This type of therapy combines unconditional laughter with yoga breathing exercises and yoga stretches, enabling patients to laugh in a different way from jokes or humour programmes. Patients in the intervention group will be divided into 2 groups of 15 patients each. A total of 12 sessions of laughter yoga will be applied to the intervention group for 6 weeks in the form of meetings via Skype application in the form of 45-minute sessions 2 times a week for 6 weeks. Laughter yoga sessions will be held every week on .......... and .......... days. Together with the patients participating in the study, the days of the laughter yoga programme will be decided to be suitable for the patients.
  Interventions: Other: laughter yoga
- Control Group (No Intervention): Laughter yoga will not be applied to patients in this group. Pre- and post-tests will be taken and observed for 6 weeks. During this period, all patients will continue to receive their routine treatment.

INTERVENTIONS:
Other: laughter yoga — Laughter yoga is a type of complementary therapy that also includes some other components, including light physical exercises. This type of therapy combines unconditional laughter with yoga breathing exercises and yoga stretching positions, enabling patients to laugh in a different way from jokes or humour programmes. Laughter yoga steps; Warm-up exercises (5-10 minutes), Deep breathing exercises (10 minutes), Childish games (10 minutes), Laughter exercises (15 minutes). During laughter yoga, laughter is achieved without any jokes, comedy or humour and supports the realisation of a sincere laughter that does not involve cognitive thinking in individuals. Laughter yoga sessions should be done at home in a quiet and calm environment by making eye contact. Laughter yoga is applied in sessions that include warm-up, breathing and laughing exercises accompanied by applause and songs. The sessions take place in groups and last 45 minutes.
  Arms: Intervention Group

SUMMARY:
The aim of this study was to evaluate the effects of laughter yoga on Fatigue, Depression-Anxiety-Stress, Sleep quality, Haematological values and Blood transfusion number in Beta Thalassemia Major patients.

DETAILED DESCRIPTION:
Beta Thalassaemia Major patients require regular transfusions at an early age due to severe anaemia. These frequent blood transfusions, which are necessary to manage anaemia in Beta Thalassaemia Major patients, cause iron overload, a major complication associated with the management of Beta Thalassaemia Major. Proximal symptoms in patients with Beta Thalassaemia Major include fatigue followed by pain, shortness of breath, palpitations, dizziness and weakness. Distal symptoms include mobility problems, sleep problems and difficulty concentrating. Mental problems such as depression and stress are also common in Beta Thalassaemia Major patients.

Material and Method: This randomised controlled study will be conducted in a total of 60 patients (30 intervention and 30 control) with the diagnosis of Beta Thalassemia Major in the Thalassemia Unit of Batman Training and Research Hospital. Patients in the intervention group will practice laughter yoga for 45 minutes 2 days a week for 6 weeks. Patient information form, Facit-Fatigue scale as primary measurement tool, Depression-Anxiety-Stress scale as secondary measurement tool, Pittsburgh sleep quality scale, haematological values of the patient and number of blood transfusions will be used to collect research data.

Implementation of the Research: Patients will be met in the thalassaemia unit and informed about the study and written consent will be obtained from patients who agree to participate in the study. The status of potential patients meeting the inclusion criteria will be determined. Depression-Anxiety-Stress Scale (DASS-42) will be applied.

Patients who fulfil the inclusion criteria will be numbered according to the order of the interview. FACIT-fatigue, Pittsburgh sleep quality scale and patient information form will be applied to the patients. Haematological values (haemoglobin, haematocrit, serum iron, serum ferritin, MCV and MCH values) and the number of erythrocyte transfusions of each patient will be obtained from the information system.

Patients will be assigned to intervention and control groups according to the randomisation list.

The primary researcher will give general information about laughter yoga to each patient in the intervention group and Skype application will be installed on the patients' smartphones for the meeting where laughter yoga sessions will be held. The phone numbers of the patients will be taken for communication, the researcher will give the number to the patients and WhatsAap groups will be created to facilitate communication. Before the laughter yoga, an information message will be sent to each patient in the intervention group and the attendance of the patients to the sessions will be checked with a follow-up chart.

Patients in the intervention group will be divided into 2 groups of 15 people each. A total of 12 sessions of laughter yoga will be applied to the intervention group for 6 weeks in the form of meetings via Skype application in the form of 45-minute sessions 2 times a week for 6 weeks. Laughter yoga sessions will be held every week on .......... and .......... days. The days of the laughter yoga programme will be decided together with the patients participating in the study, as appropriate for the patients.

At the end of the 6th week, patients in both groups will come to the thalassaemia unit. In the unit, FACIT-fatigue, Depression-Anxiety-Stress and Pittsburg sleep quality scale will be applied to the patients and haematological values and number of erythrocyte transfusions will be taken from the information system of the hospital (post-test measurements). Patients in the intervention group will be performed at least 2 days after the session to exclude the acute effect of laughter yoga.

Patients in both groups will continue to use routine treatments for 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Beta Thalassaemia major,
* Over 18 years of age,
* No hearing and communication problems,
* The one with the smartphone
* Routine treatment with iron chelators, folic acid and magnesium
* Do not have a physical problem that will prevent yoga exercises (bleeding haemorrhoids, all kinds of hernia, persistent cough, incontinence, severe back pain, hypertension, major psychiatric diseases, pregnancy, flu, epilepsy, surgery in the last 3 months, etc.)
* Depression-Anxiety-Stress scale scores of 10 and above for depression (depressed), 8 and above for anxiety (anxious), 15 and above for stress (stressed)
* Beta thalassaemia major patients who volunteered to participate in the study will be included in the study sample

Exclusion Criteria:

* Who doesn't practice laughter yoga
* Changing the treatment regime
* Patients who wish to withdraw from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The Chronic Disease Therapy-Functional Assessment of Fatigue (FACIT-Fatigue) Scale | 6 week
  The FACIT-Fatigue Scale will be used as the primary outcome measure. The Chronic Disease Therapy-Functional Assessment of Fatigue (FACIT-Fatigue) Scale is an old measure of fatigue based on classical test theory. The FACIT-Fatigue Scale consists of 13 statements measuring the fatigue experienced by patients in the last seven days. The statements in the scale consist of a Likert-type questionnaire scored between 0 and 4 and consist of 'Not at all', 'A little', 'A little', 'Quite a bit', 'Quite a lot' and 'Very much' options. The total score range of your scale is 0-52. The higher the scale score, the lower the patient's level of fatigue and vice versa. Items 1, 2, 3, 4, 4, 5, 6, 6, 9, 10, 11, 12, 13 in the scale are reverse scored, while items 7 and 8 are scored normally. It is reported that perceived fatigue is clinically severe if the score obtained from the scale is 30 and below. FACIT-F will be evaluated 2 times in total, at the beginning and at the end of the 6th week.

SECONDARY OUTCOMES:
Depression-Anxiety-Stress Scale (DASS-42) | 6 week
  The scale is 4-point Likert type and consists of 3 sub-dimensions (depression, anxiety, stress). Each sub-dimension has 14 items and there are 42 items in total in the scale. Depression items (3, 5, 10, 13, 16, 17, 21, 21, 24, 26, 31, 34, 37, 38, 42) evaluate helplessness, worthlessness, discontent, loss of interest and low energy level. Anxiety items (2, 4, 7, 9, 15, 15, 19, 20, 23, 25, 28, 30, 36, 40, 41) measure the level of muscle response, autonomic arousal, subjective and situational anxiety. Stress items (1, 6, 8, 11, 12, 14, 18, 22, 27, 29, 32, 33, 35, 39) assess the level of discomfort, difficulty relaxing, overreacting, nervous arousal, intolerance, easy upset and boredom. Depression is divided into 5 categories as remission (0-9), mild (10-13), moderate (14-20), advanced (21-27) and very advanced (28-42); anxiety remission (0-7), mild (8-9), moderate (10-14), advanced (15-19) and very advanced (20-42) and stress remission (0-14), mild (15-18), moderate (19-25), advanced (26
Pittsburgh Sleep Quality Scale (PSQS) | 6 week
  The scale includes 24 questions. Nineteen of these questions are self-assessment questions. Five questions are answered by the spouse or a friend of the individual. These five questions are used for clinical information and are not included in the scoring. Self-assessment questions include different factors related to sleep quality.
  The 18 scored items were grouped into 7 component scores. Some of the components consist of a single item, while others are obtained by grouping several items. Each item is evaluated with a score between 0 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Kıyak, Professor, Study Director — Ataturk University
Locations (1):
- Batman Training and Research Hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I want my work data to remain private

REFERENCES:
- See also: Thalassemia is an inherited blood disorder affecting hemoglobin synthesis which leads to chronic hemolysis — https://pubmed.ncbi.nlm.nih.gov/37383528/
- See also: Thalassaemia is a common inherited haematological disease. Thalassaemia major (TM) is characterised by either the lack of or reduced production of globin chains. — https://pubmed.ncbi.nlm.nih.gov/36072082/
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/36072082/ — The Effect of Happiness Training on Psychological Well-Being in Patients with Thalassaemia Major: A quasi-experimental study